CLINICAL TRIAL: NCT04375956
Title: Prospective, Non Randomized, Phase II Study on MK-3475 in Recurrent, Platinum Resistant, CPS >1 Positive Ovarian, Fallopian Tube and Primary Peritoneal Cancer Patients.
Brief Title: Study on Pembrolizumab in Recurrent, Platinum Resistant, CPS >1 Positive Ovarian, Fallopian Tube and Primary Peritoneal Cancer Patients
Acronym: MITO 27
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3094
Record Dates: First submitted 2020-04-13; First posted 2020-05-06 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg d1 q 21 iv infusion, until disease progression of disease, unacceptable toxicity or patient's refusal. Pembrolizumab will be administered for a maximum of 2 years.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Experimental

SUMMARY:
This is a single arm phase II, multicenter study evaluating Pembrolizumab in recurrent platinum resistant CPS score >1 positive ovarian, Fallopian tube and primary peritoneal cancer patients.

DETAILED DESCRIPTION:
This is a single arm, phase II, multicenter study trial evaluating Pembrolizumab in recurrent platinum resistant CPS score >1 positive ovarian, Fallopian tube and primary peritoneal cancer patients. All the eligible patients will receive Pembrolizumab 200 mg d1 q 21 iv infusion in 30 minutes, until disease progression of disease, unacceptable toxicity or patient's refusal. Pembrolizumab will be administered for a maximum of 2 years.

The primary objective of the study is to assess overall survival (OS) of patients treated with Pembrolizumab single agent.

ELIGIBILITY:
Inclusion Criteria:

1. Platinum resistant (platinum free interval 1-6 months from last platinum dose) ovarian, Fallopian tube or primary peritoneal cancer
2. CPS score>1
3. Be willing and able to provide written informed consent/assent for the trial.
4. Be >= 18 years of age on day of signing informed consent.
5. Have measurable disease or evaluable based on RECIST 1.1 (patients with only CA 125 increase without evidence of disease are not included).
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has received >2 previous CHT lines
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting
8. Has a known additional malignancy that is progressing or requires active treatment.

   Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
16. Female subjects of childbearing potential should be willing to use 2 methods of Birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
17. Patients should not be breast-feeding during treatment and for 120 days following the end of treatment
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
20. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 44 months
  The length of time from the date of the start of treatment to death

SECONDARY OUTCOMES:
Advers Events | 44 months
  The safety and tolerability of patients receiving Pembrolizumab will be assessed
Response Rate | 44 months
  The response rate will be assessed by RECIST 1.1 criteria
Progression Free Survival | 44 months
  The length of time from the start of treatment to the disease progression
Quality of life: physical impact of disease | 44 months
  Patient-reported outcomes of patients receiving pembrolizumab will be assessed utilizing the disease-related symptoms - physical (DRS-P) subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCNFACT) FACT-Ovarian Symptom Index 18 (FOSI-18) Changes and using Euro-Quality of Life 5D (eEQ-5D) tool
Quality of life: emotional impact of disease | 44 months
  Patient-reported outcomes of patients receiving pembrolizumab will be assessed utilizing the disease-related symptoms - physical (DRS-P) subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCNFACT) FACT-Ovarian Symptom Index 18 (FOSI-18) Changes and using Euro-Quality of Life 5D (eEQ-5D) tool

OTHER OUTCOMES:
CPS score | 24 months
  Correlation between different CPS score cut off and response to Pembrolizumab treatment
Concentration of Lymphoid or myeloid-derived suppression cells | 44 months
  Correlation between lymphoid or myeloid-derived suppression cells (MDSC) and response to Pembrolizumab treatment
Concentration of T-regulatory cells | 44 months
  Correlation between T-regulatory cells (T-regs) and response to Pembrolizumab treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy